CLINICAL TRIAL: NCT04925921
Title: AVAVA SR-1 Wrinkles and BPL Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AVAVA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AV-21-003
Record Dates: First submitted 2021-06-02; First posted 2021-06-14 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Wrinkle; Benign Pigmented Lesion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (Experimental): Treatment with the SR-1 Laser
  Interventions: Device: SR-1 Laser

INTERVENTIONS:
Device: SR-1 Laser — 3-4 treatments at 4-6 week intervals
  Other Names: SR-1 Skin Treatment System

SUMMARY:
This study is being conducted to evaluate the safety and efficacy of a laser called the SR-1 Skin Treatment System, or SR-1 Laser, for the treatment of wrinkles and pigmented spots. Participants will be treated with the SR-1 Laser 3 or 4 times with each treatment spaced 4-6 weeks apart. The improvement in wrinkles and pigmented spots will be evaluated 1 and 3 months after the final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Wrinkles on both sides of the face (e.g., peri-oral, peri-orbital, and cheek) scored 4-9 on the Fitzpatrick Wrinkle and Elastosis Scale
2. Willingness to have both sides of the face exposed to the SR-1 Laser.
3. Willingness to have digital photographs taken of their face and agreement with use of photographs, with their identity protected, for presentation, educational, or marketing purposes.
4. Willingness to comply with the following during the study, including the follow-up period:

   1. maintain consistent skin care regimen on treated areas
   2. cover treated areas or have very limited sun exposure and use a provided sunscreen as directed by the Investigator
   3. refrain from using systemic corticosteroids
   4. refrain from using systemic or topical skin-lightening medications or retinoids
   5. refrain from any other procedures in the treatment areas
5. Willingness and ability to comply with study instructions and return for required visits.

Exclusion Criteria:

1. Skin pathology or condition, or medication use that could interfere with evaluation of the study procedure, e.g.,

   1. Isotretinoin use within previous 6 months
   2. Surgical treatment in the target areas within previous 6 months
   3. Active vitiligo, psoriasis, or eczema, or history of these in the treatment area
2. Injection of botulinum toxin in the treatment areas within the previous 3 months.
3. Facial cosmetic procedures in the target areas within previous 6 months (e.g., laser or other energy-based device treatment, microdermabrasion, microneedling, chemical peel, injection of dermal filler).
4. Current smoker or history of smoking greater than 0.5 pack/day in past 5 years.
5. Excessive sun exposure in the previous month, or unable or unlikely to refrain from tanning or excessive sun exposure during the study.
6. Artificial tanning (e.g., tanning bed or tanning lotion/spray) in the target areas within previous 1 month or intention to use artificial tanning during the study.
7. Active localized or systemic infection, or an open wound in area being treated.
8. History of abnormal wound healing or abnormal scarring (e.g., hypertrophic or keloid).
9. History of connective tissue disease, such as lupus or scleroderma.
10. History of seizure disorders due to light.
11. Any use of medication that is known to increase sensitivity to light according to Investigator's discretion (e.g., topicals sensitive to light may be used in other areas off-face).
12. History of gold therapy.
13. History of disease stimulated by heat, such as recurrent herpes simplex or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
14. History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer. Current cancerous lesion in the treatment area.
15. Pregnancy or lactation, or intent to become pregnant within the study period.
16. Significant uncontrolled concurrent illness, such as diabetes mellitus, hypertension, or cardiovascular disease.
17. History of immunosuppression/immune deficiency disorder or currently using immunosuppressive medications.
18. Planned weight loss of greater than five pounds.
19. Facial hair in the treatment areas which would prevent evaluation of the outcome measures.
20. Current enrollment in a clinical study of any other investigational drug or device, or has received an investigational drug or been treated with an investigational device within 6 months prior to entering this study, unless the other clinical study only involves noninvasive imaging.
21. Any other physical or mental condition, or laboratory value, that would, in the professional opinion of the Investigator, potentially affect response or participation in this clinical study, or would pose an unacceptable risk to the subject.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-07-25 (Actual)

PRIMARY OUTCOMES:
Improvement in facial wrinkles | 3 months after the final treatment
  A 1 point or greater reduction in facial wrinkle severity using the Fitzpatrick Wrinkle and Elastosis Scale (FWS), as assessed, and agreed upon by at least two of three blinded independent reviewers in at least 70% of subjects as determined with a side-by-side evaluation of baseline and post-treatment photographs. The FWS scores range from 1 to 9 with lower numbers representing less severe wrinkles.

SECONDARY OUTCOMES:
Reduction of pigmentation in benign pigmented lesions (BPL) | 3 months after the final treatment
  If clinically identifiable BPL were present at baseline, a greater than 25% reduction in pigmentation of BPL (including, but not limited to, lentigos, solar lentigos, ephelides, and melasma) as assessed, and agreed upon, by at least two of three blinded independent reviewers in at least 50% of subjects as determined with a side-by-side evaluation of baseline and post-treatment photographs.
Subject satisfaction with the improvement in wrinkles | 1 and 3 months after the final treatment
  The percent of subjects satisfied with the improvement in fine lines and wrinkles in the treated areas will be assessed using a Likert scale with responses ranging from "very dissatisfied" to "very satisfied".
Subject satisfaction with the improvement in BPL | 1 and 3 months after the final treatment
  The percent of subjects satisfied with the improvement in BPL pigmentation will be assessed among subjects with clinically identifiable BPL present at baseline using a Likert scale with responses ranging from "very dissatisfied" to "very satisfied".
Tolerance of procedure | during treatment
  Subject tolerance of the procedure based on pain scores during treatment per the 1-10 Visual Analog Scale.
Adverse Events | 3 months after the final treatment
  The incidence and severity of adverse events
Overall improvement | 1 and 3 months after the final treatment
  Rate of overall improvement in facial wrinkles and BPL in the treated area(s) as assessed by the investigator using the Global Aesthetic Improvement Scale (GAIS). Wrinkles and BPL will be considered together and one overall score will be created. Scores on the GAIS range from 0 to 4 which correspond to "worsening of conditions", "no improvement in conditions", "mild improvement in conditions", "moderate improvement in conditions", and "significant improvement in conditions".

CONTACTS AND LOCATIONS:
Locations (1):
- AVAVA, Inc., Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Fitzpatrick RE, Goldman MP, Satur NM, Tope WD. Pulsed carbon dioxide laser resurfacing of photo-aged facial skin. Arch Dermatol. 1996 Apr;132(4):395-402. PMID 8629842